CLINICAL TRIAL: NCT01180998
Title: Clinical Evaluation of Two Toric Contact Lenses in Current Non-toric Lens Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Collaborators: Visioncare Research Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR-201004
Record Dates: First submitted 2010-08-11; First posted 2010-08-13 (Estimated); Results first posted 2013-12-20 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2017-06

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Spherical contact lens users (Other): Habitual spherical contact lens (non-toric lens) users tried one of two toric lenses in a daily wear modality.
  Interventions: Device: Senofilcon A Toric (AOfA); Device: Etafilcon A Toric (1DAMfA)
- Contact lens drop-outs (Other): Habitual spectacle users (for vision correction) who have failed contact lens fit and wear, tried one of two toric lenses in a daily wear modality.
  Interventions: Device: Senofilcon A Toric (AOfA); Device: Etafilcon A Toric (1DAMfA)
- Habitual Correction with Spectacles (Neophytes) (Other): Habitual spectacle lens wearers (for vision correction) who have never used or been fitted with contact lenses tried one of two toric lenses in a daily wear modality.
  Interventions: Device: Senofilcon A Toric (AOfA); Device: Etafilcon A Toric (1DAMfA)

INTERVENTIONS:
Device: Senofilcon A Toric (AOfA) — Soft toric contact lenses for astigmatism
Device: Etafilcon A Toric (1DAMfA) — Soft toric contact lenses for astigmatism

SUMMARY:
The purpose of this study is to evaluate the clinical performance, defined as successful fit, of two toric contact lenses (one daily disposable and the other daily wear reusable contact lens to correct astigmatism) in current spherical soft contact lens wearers, contact lens drop-outs, and non-users of toric contact lenses (neophytes).

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following conditions prior to inclusion in the study:

1. One of the following:

   1. Spherical contact lens user (minimum of 2 months wear, four days a week, 8 hours a day)
   2. Contact Lens drop-out (no contact lens wear in the last 6 months but wearing glasses at least four days a week,8 hours a day)
   3. Neophyte (no habitual contact lens wear except for trial fits up to 1 week, but wearing glasses at least four days a week,8 hours a day For patients not currently wearing lenses, patient should have expressed a desire to try lenses.
2. Between 16 and 60 years of age.
3. Have signed an informed consent form (documented by the investigator in the Case Report Form [CRF]).
4. Distance requirement in the range of +4.00D to -9.00D (i.e. -10.00D refractive)
5. Refractive astigmatism between -0.75D and -3.00D in both eyes.
6. Have best corrected VA of 6/9 (20/30) or better in each eye.
7. Have normal eyes with no evidence of abnormality or disease. For the purpose of this study a normal eye is defined as one having:

   1. No amblyopia.
   2. No evidence of lid abnormality or infection.
   3. No conjunctival abnormality or infection.
   4. No clinically significant slit lamp findings (i.e. stromal haze, staining, scarring, vascularisation, infiltrates or abnormal opacities).
   5. No other active ocular disease.
8. Presbyopes may be included (no monovision, no spectacles over contact lenses or bifocal glasses only)

Exclusion Criteria:

Any of the following will render a subject ineligible for inclusion:

1. Requires concurrent ocular medication.
2. Clinically significant (Grade 3 or 4) corneal stromal haze, corneal vascularisation, tarsal abnormalities, bulbar hyperaemia, limbal hyperaemia, or any other abnormality of the cornea that would contraindicate contact lens wear.
3. Corneal staining Grade 3 in more than two regions.
4. Extended wear in the last 3 months.
5. Has had any anterior ocular surgery. Has had any other ocular surgery or injury within 8 weeks immediately prior to enrollment for this study.
6. Abnormal lachrymal secretions.
7. Pre-existing ocular irritation that would preclude contact lens fitting.
8. Keratoconus or other corneal irregularity.
9. Any systemic illness which would contraindicate lens wear or the medical treatment of which would affect vision or successful lens wear.
10. Has diabetes.
11. Infectious disease (e.g., hepatitis, tuberculosis) or an immunosuppressive disease (e.g., HIV).
12. Pregnancy, lactating, or planning a pregnancy at the time of enrollment.
13. Participation in any concurrent clinical trial or in last 60 days.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2010-06-01 (Actual); Primary Completion 2010-10-01 (Actual); Study Completion 2010-10-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- United Kingdom (18):
  - Reading, Berkshire
  - Marlow, Bucks
  - Broadstone, Dorset
  - Portchester, Hampshire
  - Southsea, Hampshire
  - St Albans, Herts
  - Shanklin, Isle Of Wight
  - Rawtenstall, Lancashire
  - Hendon, London
  - Pinner, Middlesex
  - Teddington, Middlesex
  - Uxbridge, Middlesex
  - Cardiff, South Glamorgan
  - Croydon, Surrey
  - Coventry, West Midlands
  - Birmingham
  - Bristol
  - Sheffield

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited and randomized to one of two parallel arms. Three categories of subjects were recruited: spherical soft lens wearers, CL drop-outs, neophytes.
Pre-assignment Details: The data from 10 subjects was disqualified from the analysis due to subjects' ineligibility being determined after enrollment.
Groups:
- Spherical Contact Lens Users: Habitual spherical contact lens (non-toric lens) users used one of two toric lenses in a daily wear modality.
- Contact Lens Drop-outs: Habitual spectacle users (for vision correction) who have failed contact lens fit and wear, used one of two toric lenses in a daily wear modality.
- Habitual Correction With Spectacles (Neophytes): Habitual spectacle lens wearers (for vision correction) who have never used or been fitted with contact lenses used one of two toric lenses in a daily wear modality.
Period: Overall Study
Arm/Group | Spherical Contact Lens Users | Contact Lens Drop-outs | Habitual Correction With Spectacles (Neophytes)
Started | 67 | 72 | 61
Completed | 63 | 68 | 51
Not Completed | 4 | 4 | 10
Not completed — Poor Vision | 0 | 2 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Protocol Violation | 1 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Poor comfort | 3 | 0 | 4
Not completed — Poor lens handling | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are of those subjects that met the inclusion/ exclusion criteria and are enrolled and randomized to a study arm.
Groups:
- Contact Lens Drop-outs: Habitual spectacle users (for vision correction) who have failed contact lens fit and wear, and used one of two toric lenses in a daily wear modality.
- Total: Total of all reporting groups
Arm/Group | Spherical Contact Lens Users | Contact Lens Drop-outs | Habitual Correction With Spectacles (Neophytes) | Total
Number analyzed (Participants) | 67 | 72 | 61 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.6 (11.8) | 39.2 (10.0) | 32.4 (12.3) | 36.3 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 18 | 33 | 71
  Male | 47 | 54 | 28 | 129
Region of Enrollment [Number; unit: participants]
  United Kingdom | 67 | 72 | 61 | 200

OUTCOME MEASURES:

1. Primary Outcome: Overall Success in Fitting With a Toric Contact Lens
Description: Percent of subjects with success with toric lens fitting defined as meeting all of the following pre-determined criteria: 1) acceptable fit, 2) orientation stability less than or equal to 20 degree rotation, 3) binocular visual acuity (VA) within one line of spectacle VA, 4) Good, very good, or excellent overall quality of Vision, and 5) good, very, good, or excellent overall lens comfort. There was not an inferential statistical analysis conducted on this outcome. Comparison was made through the use of 95% CI's for the proportions. Therefore no statistical analysis section is included for this primary outcome.
Time Frame: 4 weeks
Population: All subjects that were dispensed a study lens except those that discontinued for non-clinical reasons.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Spherical Contact Lens Users | Contact Lens Drop-outs | Habitual Correction With Spectacles (Neophytes)
Number analyzed (Participants) | 66 | 70 | 56
percentage of participants | 80 [71 to 90] | 74 [64 to 85] | 70 [58 to 82]

2. Primary Outcome: Distance Visual Acuity
Description: Measured monocularly (each eye separately) in Snellen converted to logMAR units. The logMAR scale has a range of -0.30 to 1.00. A value of 0 or less would not require distance vision correction and a value of 0 or greater may require distance vision correction.
Time Frame: after 1 week of toric contact lens wear
Population: All subjects that were dispensed a study lens except those that discontinued for non-clinical reasons.
Measure: Least Squares Mean (Standard Error); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Spherical Contact Lens Users | Contact Lens Drop-outs | Habitual Correction With Spectacles (Neophytes)
Number analyzed (Participants) | 67 | 72 | 61
Number analyzed (eyes) | 128 | 136 | 102
logMAR
  1DAMfa Lens | -0.03 (0.01) | 0.01 (0.01) | 0.01 (0.01)
  AofA Lens | -0.01 (0.01) | 0.05 (0.02) | 0.02 (0.02)
  Total Monocular VA | -0.02 (0.01) | 0.02 (0.01) | 0.02 (0.01)

3. Primary Outcome: Distance Visual Acuity (VA)
Description: Visual Acuity is measured monocularly (each eye separately) in Snellen, the converted to logMAR units. The logMAR scale has a range of -0.30 to 1.00. A value of 0 or less would not require distance vision correction and a value of 0 or greater may require distance vision correction.
Time Frame: after 4 weeks of toric contact lens wear
Population: All subjects that were dispensed a study lens except those that discontinued for non-clinical reasons.
Measure: Least Squares Mean (Standard Error); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Spherical Contact Lens Users | Contact Lens Drop-outs | Habitual Correction With Spectacles (Neophytes)
Number analyzed (Participants) | 63 | 68 | 51
Number analyzed (eyes) | 124 | 132 | 94
logMAR
  1DAMfa Lens | -0.03 (0.01) | 0.01 (0.01) | 0.01 (0.01)
  AOfA Lens | 0.01 (0.01) | 0.04 (0.02) | 0.02 (0.02)
  Total Monocular VA | -0.02 (0.01) | 0.02 (0.01) | 0.00 (0.01)

ADVERSE EVENTS:
Groups:
- Spherical Contact Lens Users: Habitual spherical contact lens (non-toric lens) users will use one of two toric lenses in a daily wear modality.
- Contact Lens Drop-outs: Habitual spectacle users (for vision correction) who have failed contact lens fit and wear, will use one of two toric lenses in a daily wear modality.
- Habitual Correction With Spectacles (Neophytes): Habitual spectacle lens wearers (for vision correction) who have never used or been fitted with contact lenses will use one of two toric lenses in a daily wear modality.
Arm/Group | Spherical Contact Lens Users | Contact Lens Drop-outs | Habitual Correction With Spectacles (Neophytes)
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/72 | 0/61
Other Adverse Events (participants affected / at risk) | 0/67 | 0/72 | 0/61

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication required agreement and written authorization from the Sponsor.